CLINICAL TRIAL: NCT00683410
Title: A Prospective, Observational Study to Monitor Safety in Patients Who Were Administered With Pneumococcal Conjugate Vaccine, 7-valent (Prevenar) 0.5 mL by Intramuscular Injection
Brief Title: Post-Marketing Study of the Safety of Prevenar (Pneumococcal Conjugate Vaccine, 7-valent)
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 0887X-102339
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2010-11-16 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-10

CONDITIONS: Vaccines, Pneumococcal Conjugate Vaccine
MeSH Terms: interventions — Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Biological: Pneumococcal Conjugate Vaccine, 7-valent (Prevenar)

INTERVENTIONS:
Biological: Pneumococcal Conjugate Vaccine, 7-valent (Prevenar)

SUMMARY:
To collect post-marketing information on the safety of Prevenar in Filipino patients

ELIGIBILITY:
Inclusion Criteria:

* All patients from the study center who received or will receive at least one dose of Prevenar according to the approved product indication.

Exclusion Criteria:

* Previously discontinued Prevenar therapy due to safety concerns.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care
Sampling Method: Non-Probability Sample
Enrollment: 3366 (Actual)
Dates: Start 2007-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- City of Muntinlupa, Philippines

RESULTS

PARTICIPANT FLOW:
Groups:
- Prevenar 7v: Pneumococcal conjugate vaccine, 7-valent, 0.5 mL intramuscular injection
Period: Overall Study
Arm/Group | Prevenar 7v
Started | 3366
Vaccinated Dose 1 | 3240
Vaccinated Dose 2 | 1623
Vaccinated Dose 3 | 817
Vaccinated Dose 4 | 175
Completed | 3366
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prevenar 7v
Number analyzed (Participants) | 3366
Age Continuous [Mean (Standard Deviation); unit: weeks] | 43.6 (50.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1576
  Male | 1790

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Spontaneous Adverse Events
Time Frame: 30 days post injection up to 3 years
Population: Safety Analysis set - all participants who received at least one dose of Prevenar
Measure: Number; unit: Participants
Arm/Group | Prevenar 7v
Number analyzed (Participants) | 3366
Participants | 91

ADVERSE EVENTS:
Time Frame: 30 days following each vaccination
Arm/Group | Prevenar 7v
Serious Adverse Events (participants affected / at risk) | 3/3366
Other Adverse Events (participants affected / at risk) | 88/3366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevenar 7v (N=3366)
Pyrexia (General disorders) | 1
Convulsion (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevenar 7v (N=3366)
Diarrhoea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Feeling abnormal (General disorders) | 1
Injection site swelling (General disorders) | 3
Irritability (General disorders) | 1
Lethargy (General disorders) | 1
Pyrexia (General disorders) | 36
Exanthema subitum (Infections and infestations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Febrile convulsion (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 7
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 7
Bronchitis acute (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Infantile asthma (Respiratory, thoracic and mediastinal disorders) | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 8
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 23
Viral rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Rash pustular (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.